CLINICAL TRIAL: NCT00164437
Title: CD-ROM Intervention for Prostate Cancer Screening
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of Colorado, Denver (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: CDC-NCCDPHP-4020; U48/CCU815787
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-09

CONDITIONS: Prostate Cancer
Keywords: screening; community healt education; decision making; computer-assisted decision making
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Behavioral: educational CD-ROM

SUMMARY:
The study populations consist of a sample of the patient population (men aged 40-79 years) of a large, group model HMO and a community sample of men age 50-79. Follow-up interviews of men randomly assigned to the intervention and control groups are being conducted by telephone to assess issues related to prostate cancer screening and the men's use of the CD-Rom educational intervention.

DETAILED DESCRIPTION:
The study populations consist of a sample of the patient population (men aged 40-79 years) of a large, group model HMO and a community sample of men age 50-79. Follow-up interviews of men randomly assigned to the intervention and control groups are being conducted by telephone to assess issues related to prostate cancer screening and the men's use of the CD-Rom educational intervention. Preliminary results are available for the first 1304 follow-up interviews (interim response rate = 26%). Of 554 men randomized to receive the CD-ROM, 227 (41%) reported receiving the CD-ROM, and 78 (14%) used it in a computer. About 51% of these 78 men used the CD-ROM once only, while 42% used it twice, and 27% shared it with someone else. Most users reported learning some (44%) or a great deal (46%) of new information from the CD-ROM, and most reported that it helped them organize their thoughts about screening somewhat (44%) or a great deal (28%). About 19% indicated that the CD-ROM increased their uncertainty somewhat or a great deal about whether or not they want to be screened, 30% reported that the CD-ROM changed their feelings about whether or not they want to be screened somewhat, and 12% reported that it changed their feelings a great deal. Men who used the CD-ROM had higher education, higher income, higher levels of computer usage, and were more likely to have previously had a PSA test compared to non-users. No other subject characteristics were significantly related to use. Using randomized group assignment in an "intention to treat" analysis, prostate cancer knowledge was significantly higher in the intervention group; there were no differences between study groups in decisional conflict or realistic expectations. However, when comparing those who did and did not use the CD-ROM using multiple regression analysis and controlling for differences in age, race, education, income, insurance status, previous receipt of prostate cancer screening, and computer usage, use of the CD-ROM was significantly associated with higher prostate cancer related knowledge, lower decisional conflict, and more realistic expectations about risk of dying from prostate cancer. After controlling for differences between users and non-users we found evidence that the CD-ROM was effective in reducing decisional conflict, and increasing knowledge and realistic expectations related to prostate cancer screening.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* prostate cancer

Min Age: 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 554
Dates: Start 2002-09; Study Completion 2004-09

PRIMARY OUTCOMES:
prostate cancer knowledge,
ability to make an informed decision about prostate cancer screning,
decisional conflict,
realistic expectations

SECONDARY OUTCOMES:
costs

CONTACTS AND LOCATIONS:
Overall Officials: Lori A. Crane, PhD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Health Sciences Center, Denver, Colorado, United States